CLINICAL TRIAL: NCT03373747
Title: Reliability Intra and Inter-evaluators and Physiological Analysis of an Isometric Test of Localized Muscular Fatigue
Brief Title: Reliability and Physiological Analysis of an Isometric Test of Localized Muscular Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Larissa Rodrigues Souto, Principal Investigator, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2016/11785-7
Record Dates: First submitted 2017-11-21; First posted 2017-12-14 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reliability of IET (Experimental): In phase 1, the first of familiarization is to the participants understand the test and familiarize with the equipment after 24 to 48 hours, the participants will do the test applied twice at the same day with 10 minutes of rest. For realization of the IET the participants will be instructe to make the maximum effort as possible and mantain until they can't resiste. After one week the retest session will be doing. The order between the evaluators will be changed in the test and retest sessions.
  Interventions: Diagnostic Test: Reliability of IET
- Physiological analysis of IET (Experimental): In phase 2, the participants will be submitted two sessions, familiarization session and test session. In the test session there is be two teste applied in the same day with approximately 20 minutes of rest. In the first test, thers is gas analysis during all the test until seven minutes after the test and blood lactat concentrate will be colected before the test with 10 minutes of rest, immediately after the teste and in the first, in the third, fifth and seventh minutes after the test. In the second test will be assess the muscular activation porcentage of lateral vastus muscle by means of twitch interpolation technique there is be performe before and after the test.
  Interventions: Diagnostic Test: Physiological analysis of IET

INTERVENTIONS:
Diagnostic Test: Reliability of IET — The participants will be do three sessions: familiarization, test and retest to assess the reliability inter and intra rater of the test.
  Arms: Reliability of IET
Diagnostic Test: Physiological analysis of IET — The participants will be submitted two sessions, familiarization session and test session. In the test session there will be the physiological analysis by means of gas analysis, blood lactate concentrate and activation muscular percentage.
  Arms: Physiological analysis of IET

SUMMARY:
Introduction: The isokinetic dynamometer, considered a gold standard tool for physical evaluation, is widely used in studies that aim to evaluate the reliability and reproducibility of localized muscular endurance (LME) tests. However, such tests may not represent full LME by fixing time or number of replicates. Therefore, it is relevant to construct a test that respects the actual capacity of each subject to withstand fatigue and to submit such a test to validation, as well as to physiological analysis.

Research objectives: To assess the inter- and intra-rater reliability of a localized isometric endurance test (IET) on the isokinetic dynamometer and to establish the metabolic demand required during the test.

Design: Reliability study with test-reteste dynamic.

Participants and Setting: After fulfilling the eligibility criteria, eighty-eight male participants will participate in the study.

Procedure: In phase 1 forty-eight participants will submitted to reliability of the IET within three sessions: familiarization session, test session and retest sessio. In phase 2 forty participants will be submitted the metabolic demand required during the IET will be analyzed by means of gas analysis, blood lactat concetrate and muscular activation percentage.

Intervention: isometric endurance teste.

Measurements: The measurements include time of execution of test, work of test, physiological and psychological outcomes.

DETAILED DESCRIPTION:
Introduction: The isokinetic dynamometer, considered a gold standard tool for physical evaluation, is widely used in studies that aim to evaluate the reliability and reproducibility of localized muscular endurance (LME) tests. However, such tests may not represent full LME by fixing time or number of replicates. Therefore, it is relevant to construct a test that respects the actual capacity of each subject to withstand fatigue and to submit such a test to validation, as well as to physiological analysis.

Research objectives: To assess the inter- and intra-rater reliability of a localized isometric endurance test (IET) on the isokinetic dynamometer and to establish the metabolic demand required during the test.

Design: Reliability study with test-reteste dynamic.

Participants and Setting: After fulfilling the eligibility criteria, eighty-eight male participants will participate in the study. The inclusion criteria include: healthy male, aged between 18-30 years who agree to participate in the study. Participants with the following will be excluded from the study: presence of anemia, inflammation, being sick, training or physical activity at least 24 hours prior the application of the test, being influenced in some way by test information, do not understand the teste and occurrence of musculoskeletal injury during the study.

Procedure: In phase 1 forty-eight participants will submitted to reliability of the IET within three sessions: familiarization session, test session and retest sessio. In phase 2 forty participants will be submitted the metabolic demand required during the IET will be analyzed by means of gas analysis, blood lactat concetrate and muscular activation percentage.

Intervention: This is a test that was developed by the Laboratory of Sports Physiotherapy of FCT/UNESP - Presidente Prudente. The test will be performed on the Biodex System Pro 4 isokinetic dynamometer (Biodex Medical System, Shirley-NY, USA). At first, participants will be be positioned and fixed on the device itself by their trunk, hips, thighs and by the distal region of the assessed lower limb (dominant). The protocol is composed by a 10 knee flexo-extension warm up at the speed of 330º/s, respecting the amplitude of 90º, then a 30 second isometric contraction from 50% to 60% of the maximum participant effort, according to the Effort Perception Scale. The test starts after two minutes of rest. So that it can take place, participants will be instructed to make as much effort as possible, according to the same scale, for as long as possible, until they can't keep muscle contraction no longer. To stimulate participants, evaluators will offer verbal motivation and they will follow a monitor, coupled to the device, which offers the power generation line which works as a visual feedback during all test long.

In phase 1, the first of familiarization is to the participants understand the test and familiarize with the equipment after 24 to 48 hours, the participants will do the test applied twice at the same day with 10 minutes of rest. For realization of the IET the participants will be instructe to make the maximum effort as possible and mantain until they can't resiste. After one week the retest session will be doing. The order between the evaluators will be changed in the test and retest sessions. In phase 2, the participants will be submitted two sessions, familiarization session and test session. In the test session there is be two teste applied in the same day with approximately 20 minutes of rest. In the first test, thers is gas analysis during all the test until seven minutes after the test and blood lactat concentrate will be colected before the test with 10 minutes of rest, immediately after the teste and in the first, in the third, fifth and seventh minutes after the test. In the second test will be assess the muscular activation porcentage of lateral vastus muscle by means of twitch interpolation technique there is be performe before and after the test.

Measurements: The measurements include time of execution of test (in seconds), work of test (in N.m), physiological (gas analysis, blood lactate concentration, muscular activation percentage) and psychological outcomes (Psychological Questionnaire, Work Ability Index Questionnaire, Perceived Stress Scale, The Bergen Insomnia Scale, Need for Recovery Scale, The Borg Scale, The Borg CR10 Scale, The Effort Perception Scale and Recovery Perception Scale) and clinical outcomes (heart rate).

Analysis: To analyse the normality will be used Shapiro Wilk test. For analysis of reliability test-retest will be used the intraclasse correlation coefficient (ICC), with confidence interval of 95% to reliability relative. To assess the reliability absolute the typical error and coefficient of variation will be done. The paired test t will be do to verify diferences n the mean of the groups. The psychological outcomes wiil be done with correlation and linear regression as well the physiologica outcomes. A significance level of 5% will be assumed for all statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (self-report);
* Male gender;
* Aged between 18-30 years;
* Agreement to participate through signed statement of informed

Exclusion Criteria:

* Being sick;
* Training or physical activity at least 24 hours priot to the application test;
* Being influenced in some way by test information;
* Do not understand the test;
* Inflammatory process;
* Cardiovascular disease;
* Episode of musculo-tendinous or osteoarticular lesion in the lower limbs and/or spine in the last seix months;

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
The time of execution of the test | 45 seconds after the beginning of the test
  This outcome will be assessed in seconds during execution of the test

SECONDARY OUTCOMES:
The work of the test | day 2 and day 7
  This outcome will be assessed in Newton.meter (N.m) during execution of the test
Oxygen consumption - gas analysis | Second phase during all the test
  Gas analysis will be measured during the test and after seven minutes of the same (VO2000, MedGraphics, Minnesota, USA).
Blood lactate concentration | Second phase, 10 minutes of rest before the test and immediately after the test and in the third, fifth and seven minutes after the test
  The blood lactate concentration will be collected in the 10 minutes of rest before the test and immediately after the test and in the third, fifth and seven minutes after the test
Muscular activation percentage | Day 2
  The muscular activation percentage will be assessed by means of twitch interpolation technique ( current generator - Quark)
Psychological Questionnaire | Day 2 and day 7
  Participants will be instructed to mark with a dash, on a 10 centimeters analogical visual scale in between two extremes, in which zero means "non-existent" and 10 "very intense" to each classification
Work Ability Index Questionnaire | Day 1
  This questionnaire consists in seven indicators, which provide a score between seven and 49, in which the highest the scores the better. These indicators evaluate occupational wellness, providing subjective estimation about work capacity, including the ability to perform work tasks in relation to demands, health and mental resources
Perceived Stress Scale | Day 1
  This scale is intended to document participants' related stress on the previous month. Items evaluate the degree to which people find life unpredictable, uncontrollable or overloaded. This scale evaluates overall beliefs about perceived stress, without the providence of any specific event lists in life to the subjects, allowing these scores not to be biased by the event content or difference of previous life experience
Bergen Insomnia Scale | Day 1
  This scale is intended to evaluate participants' sleep and tiredness, which consists in six questions about sleep issues in the previous month. Questions are about (1) problems initiating sleep, (2) awakening from sleep, (3) early morning awakening, (4) not feeling adequately rested, (5) experiencing daytime impairment and (6) being dissatisfied with sleep. To each question participants will answer on a zero to seven days a week scale. The quantity of days will be calculated based on the average of the answers to these six questions, in order to obtain an overall sleep problems score
Need for Recovery Scale | Day 7
  This is an 11 item scale which aims to evaluate work fatigue symptoms, related to a series of emotional, cognitive and behavioral aspects characterized as temporary overload feelings, irritability, social seclusion, lack of energy for new efforts and performance reduction
Borg Scale | Day 7
  Participants' physical effort perception will also be measured by the Borg Scale, which will be used to correlate with heart rate values. After the completion of IET participants willl answer the following question: "How much exertion did you experience during the test? ". This scale has 15 possible answers, ranging from six to 20, represented respectively from "not exertion at all" to "maximal exertion".
Borg CR10 Scale | Day 7
  Participants' physical effort perception will be measured by The Borg CR10 Scale. After the IET application participants will answer the following question: "How much exertion did you experience during the test? ". This scale has 16 possible answers which vary from zero to 10 represented respectively from no effort to maximum effort.
Effort Perception Scale | Day 1, day 2 and day 7
  The effort perception will be evaluated by the Effort Perception Scale, with values between 0 and 10, 0 being correspondent to no effort at all (rest) and 10, to maximum effort
Recovery Perception Scale | Day 1, day 2 and day 7
  The perceived recovery of the dominant lower limb will be assessed by means of the Effort Perception Scale, which consists of a 10-point Likert Scale, in which 1 means no recovery and 10, completely recovered
Heart Rate | Day 2 and day 7
  The heart rate caption will take place using a cardio frequency meter (Polar electro, Oy Kempele, Finland - V800 model)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Pastre, PhD, Principal Investigator — Univ Estadual Paulista
Locations (2):
- Brazil (2):
  - Larissa Rodrigues Larissa Rodrigues Souto, Presidente Prudente, São Paulo
  - Larissa Rodrigues Souto, Presidente Prudente, São Paulo

IPD SHARING:
Plan to Share IPD: No